CLINICAL TRIAL: NCT00664053
Title: Effects of DHEA/Exercise on Bone, Muscle and Balance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Aeronautics and Space Administration (NASA) (U.S. Federal Agency)
Collaborators: University of Connecticut (Other)
Responsible Party: Anne Kenny, MD, Associate Professor of Medicine, University of Connecticut Center on Aging
Organization: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: AG0099; NNG04GK63G
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2008-04-29 (Estimated); Status verified 2008-04

CONDITIONS: Osteoporosis; Frailty
Keywords: bone mineral density; bone turnover markers; strength; balance
MeSH Terms: conditions — Osteoporosis; Frailty | interventions — Dehydroepiandrosterone; Yoga; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): DHEA and Yoga
  Interventions: Dietary Supplement: DHEA; Behavioral: Yoga
- 2 (Active Comparator): DHEA and exercise
  Interventions: Dietary Supplement: DHEA; Behavioral: Aerobics
- 3 (Active Comparator): Placebo and Yoga
  Interventions: Behavioral: Yoga; Dietary Supplement: Placebo
- 4 (Placebo Comparator): Placebo and exercise
  Interventions: Dietary Supplement: Placebo; Behavioral: Aerobics

INTERVENTIONS:
Dietary Supplement: DHEA — 50mg daily for 6 months
  Other Names: Dehydroepiandrosterone
  Arms: 1; 2
Behavioral: Yoga — 2 sessions per week for 6 months
  Arms: 1; 3
Dietary Supplement: Placebo — Placebo supplement every day for 6 months
  Arms: 3; 4
Behavioral: Aerobics — Walking/chair aerobics program 2 sessions per week for 6 months
  Arms: 2; 4

SUMMARY:
The purpose of this study is to examine whether muscle strength and balance will improve in women with frailty selected for dehydroepiandrosterone sulfate (DHEAS) levels below 550 ng/dl treated with DHEAS supplementation and Hatha yoga. Investigators believe the effects of both treatments will improve outcomes more than either treatment alone and may be additive; in addition, lean body mass, skeletal muscle mass, markers of bone turnover and physical performance will improve following treatment with DHEA and/or yoga.

DETAILED DESCRIPTION:
Dehydroepiandrosterone (DHEAS) and yoga may mitigate or reverse the effects of aging and frailty on bone, muscle and balance loss. The mechanism of the effects may be direct - working through androgen or estrogen receptors in bone, muscle or brain. Or the effects may be indirect, countering effects of the stress response.

The specific aims of this study are:

1. To determine the effects of dehydroepiandrosterone sulfate (DHEAS) supplementation and/or Hatha yoga on muscle strength, balance, body composition and physical performance measures over 6 months in women with osteopenia and some degree of frailty
2. To determine the effect of dehydroepiandrosterone sulfate (DHEAS) supplementation and/or Hatha yoga on function (physical and cognitive), bone metabolism, and cardiovascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Women over age 65 years
* Bone mineral density t-score less than -1
* At least one of the five components of the frailty phenotype (low hand grip strength, low walking speed, low physical activity, weight loss or sense of exhaustion)
* DHEAS levels less than 550 ng/dl
* Able to come or be brought to the University of Connecticut Health Center (UCHC) for outpatient visits
* Mammogram within the preceding 12 months

Exclusion Criteria:

* Disease or medication known to affect bone or muscle metabolism (i.e., Paget's disease, osteomalacia or 25OHD level less than 10 ng/dl, hyperparathyroidism: current use of corticosteroids, calcitonin, heparin, phenytoin, phenobarbital, methotrexate, bisphosphonates, calcitonin, selective estrogen receptor modulator or PTH)
* Use of androgen or estrogen in the preceding year
* Use of psychiatric medications including antipsychotic medications and SSRI
* Metastatic or advanced cancer (other than skin cancer)
* History of breast cancer
* Active cardiac ischemia by history of angina or myocardial infarction in the preceding 6 months

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 99 (Actual)
Dates: Start 2004-10; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Muscle strength, bone turnover markers | baseline, 3 month and 6 months

SECONDARY OUTCOMES:
Changes in activities of daily living, cognitive and emotional function | baseline and 6 months
Laboratory tests to measure factors that may reflect or influence changes in bone metabolism | baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Anne Kenny, MD, Principal Investigator — University of Connecticut Center on Aging
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

REFERENCES:
- [Background] von Muhlen D, Laughlin GA, Kritz-Silverstein D, Bergstrom J, Bettencourt R. Effect of dehydroepiandrosterone supplementation on bone mineral density, bone markers, and body composition in older adults: the DAWN trial. Osteoporos Int. 2008 May;19(5):699-707. doi: 10.1007/s00198-007-0520-z. Epub 2007 Dec 15. PMID 18084691
- [Background] Wang YD, Wang L, Li DJ, Wang WJ. Dehydroepiandrosterone inhibited the bone resorption through the upregulation of OPG/RANKL. Cell Mol Immunol. 2006 Feb;3(1):41-5. PMID 16549048
- [Background] Greendale GA, McDivit A, Carpenter A, Seeger L, Huang MH. Yoga for women with hyperkyphosis: results of a pilot study. Am J Public Health. 2002 Oct;92(10):1611-4. doi: 10.2105/ajph.92.10.1611. No abstract available. PMID 12356608
- [Derived] Kenny AM, Boxer RS, Kleppinger A, Brindisi J, Feinn R, Burleson JA. Dehydroepiandrosterone combined with exercise improves muscle strength and physical function in frail older women. J Am Geriatr Soc. 2010 Sep;58(9):1707-14. doi: 10.1111/j.1532-5415.2010.03019.x. PMID 20863330